CLINICAL TRIAL: NCT07103226
Title: Analysis of Hyperthermia as an Adjunctive Treatment to Evidence-based Clinical Intervention in Subjects With Plantar Fasciitis: a Double-blind Randomized Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Manuel González-Sánchez, Principal Investigator, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 139/2025
Record Dates: First submitted 2025-07-25; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Plantar Fascia; Hyperthermia
MeSH Terms: conditions — Hyperthermia | interventions — Diathermy; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hyperthermia 2 times per week (Experimental)
  Interventions: Radiation: Hyperthermia; Other: Physical Exercise; Other: Stretching; Other: Orthopedic insole
- Hyperthermia 3 times per week (Experimental)
  Interventions: Radiation: Hyperthermia; Other: Physical Exercise; Other: Stretching; Other: Orthopedic insole
- Non-hyperthermia 2 times per week (Experimental)
  Interventions: Other: Physical Exercise; Other: Stretching; Other: Orthopedic insole
- Non-hyperthermia 3 times per week (Experimental)
  Interventions: Other: Physical Exercise; Other: Stretching; Other: Orthopedic insole

INTERVENTIONS:
Radiation: Hyperthermia — Hyperthermia will be applied for a period of 15 to 20 minutes in the area to be treated, maintaining a thermal sensation of gentle heat for the patient and accompanied by active-assisted or passive mobilization of the structures adjacent to the plantar fascia.
  Arms: Hyperthermia 2 times per week; Hyperthermia 3 times per week
Other: Physical Exercise — The therapeutic physical exercise focused on the flexor muscles of the foot will consist of 3 periods of isometric contraction of 15 seconds, with a rest period of 30 seconds, varying the number of repetitions from 3 to 5 depending on the patient's symptoms.
Other: Stretching — The plantar fascia stretch will be performed with the patient in the supine position. Maximum dorsiflexion will be achieved, and the lower limb will be elevated with the knee extended as tolerated. This procedure will be performed three times in a row for 30 seconds, with a 1-minute rest between each stretch.
Other: Orthopedic insole — Imposition of an orthopedic insole

SUMMARY:
This project aims to analyze the use of hyperthermia within a treatment protocol for plantar fasciitis, as well as to determine the difference between two and three sessions per week. Study participants will be divided into four intervention groups: the first will receive two sessions per week for a period of six months, while the second will receive three sessions per week for the same period. The treatment protocol will consist of therapeutic physical exercise focused on the foot muscles and stretching the plantar fascia and posterior chain, hyperthermia on the plantar fascia insertion area in the calcaneus and adjacent areas, and the use of an orthotic insole used for walking. The third and fourth intervention groups will receive the same treatment as mentioned above, but without hyperthermia. The third group will receive three sessions per week, while the second group will receive two sessions per week. Two different types of measurement variables will be used: objective variables will be used to measure local pain using an algometer, assess ankle joint range of motion, and use ultrasound imaging techniques. Subjective variables will also be used through validated questionnaires, which will address physical activity, perceived functional limitations in patients with lower limb pathologies, lower limb functional assessment, and a visual analogue scale for pain perception.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis confirmed by performing an ultrasonography of Plantar Fascitis
* Have not yet received physiotherapy treatment.

Exclusion Criteria:

* Have undergone surgery.
* Those who refuse to participate in this study.
* Patients with muscle atrophy due to plantar fasciitis.
* Medical conditions that are contraindications for hyperthermia therapy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
FOOT AND ANKLE ABILITY MEASURE (FAAM) | Baseline and up to one year
  This instrument is based on the subjective assessment of physical function and activities of daily living in patients with musculoskeletal disorders of the lower limb. It consists of 29 items, divided into two subscales: activities of daily living (21 items) and sports activities (8 items). Each question can be scored on a scale from 4 (no difficulty) to 0 (total inability to perform the activity in question). The maximum score is 84 for the activities of daily living subscale and 32 for sports activities, representing full functionality. The Spanish version has been shown to be correctly translated from its original version and to present a correct structure, internal consistency, reliability, correlation between the total items and between items, and validity.
LOWER EXTREMITY FUNCTIONAL SCALE (LEFS) | Baseline and up to one year
  This questionnaire assesses perceived functionality in patients with a musculoskeletal problem in the lower limb. It consists of 20 questions, each of which is scored by the patient, ranging from 0 (extreme difficulty or inability to perform the activity) to 4 (no difficulty). The maximum score is 80 (no functional limitations), and the minimum score of 0 indicates extreme limitation. The Spanish adaptation has demonstrated similar values to the English version in the areas of internal consistency, reliability, structure, and error.
International Physical Activity Questionnaire (IPAQ) | Baseline and up to one year
  This instrument is designed to measure physical activity levels in an adult population and can serve as a reference for making recommendations regarding physical activity. It comes in two versions: the long version with 31 items (IPAQ-LF) and the short version with 9 items (IPAQ-SF). The short version, which will be used in this study as recommended by the authors, measures activity at four intensity levels, ranging from 1 (vigorous-intensity activity) to 4 (sedentary). It has very good reliability (r=0.8).
Visual Analogue Scale (VAS) | Baseline and up to one year
  It consists of an 11-point numerical scale, ranging from 0 (no pain) to 10 (maximum pain intensity), which serves as a quantification for measuring pain intensity. It has moderate to good reliability.
PRESSURE PAIN THRESHOLD (PPT) | Baseline and up to one year
  Pressure Pain Threshold (PPT) has proven to be a reliable method for measuring pain intensity in patients with plantar fasciitis. To perform this test, the patient is placed prone, and the most painful point under the heel is palpated. Once located, a portable mechanical pressure algometer is used, increasing pressure at a rate of 30 kPa/s. The patient is provided with a portable switch that they can activate when the session changes from pressure to pain. This procedure is repeated three times, with a 30-second rest period between tests.
WEIGHT-BEARING LUNGE TEST (WBLT) | Baseline and up to one year
  The Weight-Bearing Lunge Test (WBLT) is a reliable method for measuring ankle joint range of motion by measuring the maximum anterior displacement of the tibia on the talus in a weight-bearing position. The patient stands facing a wall with their fingers on the wall for balance and the healthy limb 30 centimeters behind the affected limb. The affected foot is placed parallel to a tape measure with the knee perpendicular to the wall, with the foot remaining in full contact with the floor. The patient is asked to touch the wall with their knee, without lifting their heel from the floor, doing this four times: the first attempt is to measure the distance from the wall, and the remaining three are used as measurements, with the average being recorded.
Ultrasonography | Baseline and up to one year
  Ultrasound imaging is an excellent noninvasive method for analyzing foot structures, including the plantar fascia. To do this, the patient is placed prone, and the transducer is positioned on the plantar surface of the heel, pointing toward the second toe, to assess the insertion of the plantar fascia into the medial tuberosity of the calcaneus. Subsequently, using the ultrasound software, three successive measurements of plantar fascia thickness are taken, first on the symptomatic foot and then on the contralateral foot. This measurement has proven to be a reliable method for assessing the plantar fascia.